CLINICAL TRIAL: NCT03607630
Title: Can Imagination Change Upsetting Memories of Trauma?
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: South London and the Maudsley NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18/LO/0684
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-06

CONDITIONS: Psychosis
Keywords: Imagery rescripting; case series; ImRs; Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Multiple Baseline Case Series - randomization for how long participants wait pre-intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waiting Pre-Intervention Control (No Intervention): Participant completes measures for 1-3 weeks (randomly chosen) before they complete the intervention. Participants act as their own controls
- Imagery Rescripting (Experimental): 3 Sessions of Imagery Rescripting
  Interventions: Other: Imagery Rescripting

INTERVENTIONS:
Other: Imagery Rescripting — psychological therapy
  Arms: Imagery Rescripting

SUMMARY:
Research suggests that imagination is a powerful tool to change images inside our heads (e.g. memories) and make them less upsetting. It is thought that this occurs through changing the meaning attached to the memory (e.g. I am weak), therefore making it less upsetting to remember.

Research has also linked some people's experience of psychosis to distressing trauma memories. Despite this, little is known about whether using imagination to change memories is helpful for people with psychosis. This project will look at whether a talking therapy that uses imagination to change trauma memories helps people with psychosis. This project will specifically look at whether this therapy helps; change the meaning linked to memory, make the memory less upsetting and frequent, and increase sense of control over the memory.

This project will recruit six to twelve people with psychosis. Participants will be recruited from services within South London and the Maudsley NHS Foundation Trust's Psychosis Clinical Academic Group. Participants will first be interviewed about their posttraumatic stress difficulties, experiences of psychosis, mental health, and wellbeing. In this appointment, participants will also identify a traumatic memory to focus on during the talking therapy. Four questions about the trauma memory will be asked every day for the remainder of the project.

Participants will then wait between one to three weeks before they receive three therapy sessions. Comparing participants to themselves for different periods of time makes sure that their memories do not become less upsetting over time, without therapy.

After therapy, participants will continue daily measures for two weeks, with an appointment in the middle (i.e. one week post therapy). This appointment will include questions about posttraumatic stress difficulties, wellbeing and satisfaction with therapy. Participation will last between 6-8 weeks. Participants will be reimbursed for their time

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Schizophrenia-spectrum disorder or mood disorder with psychotic features
* Able to identify an intrusive traumatic memory occurring at least twice in the past week, as assessed by the Post Traumatic Stress Diagnostic Scale.
* Sufficient English to participate in the project

Exclusion Criteria:

* Concurrent trauma-focused psychological therapy
* Primary diagnosis of learning disability, substance use or organic disorder
* Acute suicide risk
* Lack of capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-03 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Daily Ratings measuring change in Index Memory throughout the project | Daily throughout the project, up to 8 weeks
  Change in participant's conviction in the distressing appraisal, frequency, distress, and sense of control associated with the memory

SECONDARY OUTCOMES:
Psychotic Symptom Rating Scales (PSYRATS; Haddock, McCarron, Tarrier, & Faragher, 1999) | First week at the initial assessment
  The PSYRATS was developed to measure dimensions of delusional beliefs (6 item Delusions Scale) and auditory hallucinations (11 item Auditory Hallucination Scale). The six items on the auditory hallucination sub-scale consists of items such as negative content, frequency, loudness, intensity and amount of distress and degree of disruption and control. The six-item delusion subscale consists of items such as duration and amount of pre-occupation, intensity and amount of distress and disruption, and degree of conviction. All items are rated on a five-point scale of increasing severity (0= No problem to 4 = Maximum severity). The PSYRATS has been shown to have good validity and reliability, with sensitivity to change (Haddock et al., 1999). This study will use the PSYRATS to describe the study sample.
Change in Wellbeing through 'The Warwick-Edinburgh Mental Well-being Scale' (WEMWBS; Tennant et al, 2007) | First week at Initial assessment and 1 week post therapy
  The WEMWBS assessed wellbeing on 14 items rated on a 5-point Likert scale, ranging from "none of the time" to "all of the time". A total score ranging from 14-70 is calculated. Higher scores indicate higher levels of mental wellbeing. WEWBS shows high reliability, low social desirability, and confirmatory factor analysis supported the single-factor hypothesis (Tennant et al., 2007). It also shows high correlations with other well-being scales and low to moderate positive correlation with overall health (Tennant et al., 2007).
Change in PTSD symptoms through 'The Posttraumatic Diagnostic Scale for DSM-5' (PDS-5; Foa et al., 2016) | First week at Initial assessment and 1 week post therapy
  a 49-item self-report measure including all DSM-IV symptom criteria. 20 of these items asks participants to rate symptoms, and two questions relate to distress and interference. It has high face validity, internal consistency and reliability (Foa et al., 2016). This study will use the symptom section assessed over the past week, in order to measure change over time.
Mini-Trauma and Life Events Checklist (mini-TALE; Hardy et al, in prep) | First week at Initial Assessment
  a brief measure of trauma history, focusing on victimisation events with a general probe for other significant events experienced. It includes 5 items, each rated for occurrence, frequency, and age of occurrence.
Semi-Structured interview (adapted from Hackmann, Clark ,& McManus's (2000) work on social phobia) | First Week at Initial Assessment
  adapted from Hackmann, Clark, & McManus's (2000) work on social phobia, also used in Ison et al. (2014). This consists of a series of standardised questions asking clients to identify an index intrusive traumatic memory. The dimensions of this index memory will be assessed during the interview, including; the associated negative appraisal, intrusion frequency, associated distress and control over the memory. A visual analogue scale ranging from 0 to 10 will be used.
Credibility and Expectancy Questionnaire (CEQ; Borkovec & Nau, 1972) | First session of therapy, this may be at week 2, 3 or 4, depending upon baseline waitlist time
  item self-report instrument that measures treatment credibility, and client expectancy for improvement. The CEQ has high internal consistency (a = 0.79-0.90). Retest reliability is r = 0.82 for the expectancy factor and r = 0.75 for the credibility factor (Devilly & Borkovec, 2000). The first four items are rated based on cognitive appraisal of the treatment (e.g. At this point, how successfully do you think this treatment will be in reducing your symptoms?), whereas the last two items are rated based on feelings about the treatment. To reduce demand characteristics, client forms will be sealed in an envelope upon completion, and clients will be told that the therapist will only see the forms after they have finished participation.
Client Satisfaction Questionnaire (CSQ-8; Larsen et al, 1979) | One week Post intervention
  an eight-item version, to evaluate patient satisfaction. The sum of the responses to the CSQ-8 ranges from 8 to 32, with higher scores indicating greater satisfaction. The CSQ-8 has demonstrated high internal consistency across a large number of studies (Attkisson & Greenfield, 1999).

CONTACTS AND LOCATIONS:
Locations (1):
- South London and the Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data will be anonymised. Participant data will only be linked with their participating documents with the research participant. This data will not be shared.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03607630/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03607630/ICF_001.pdf